CLINICAL TRIAL: NCT06358365
Title: Evaluation of the Safety & Performance of the Aquapass -Medical Device, for Enhancing Fluid Transfer Through the Skin, by Increased Sweat Rate, on Hemodialysis Patients
Brief Title: Enhancing Fluid Transfer Through the Skin, by Increased Sweat Rate, on Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AquaPass Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQP-DCL-026
Record Dates: First submitted 2024-01-15; First posted 2024-04-10 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adult patients undergoing regular hemodialysis (Experimental): This study will be a crossover study with one center and an open label design. Patients who sign the informed consent form and meet the inclusion and exclusion criteria will undergo a 2-hour acclimatization period to verify their ability to adhere to the AquaPass procedure. Once enrolled, patients will undergo a 3-week observation period where they will continue with their regular hemodialysis treatment with no changes. Study endpoint parameters will be assessed during this observation period and used as a control group. After the observation period, patients will undergo the AquaPass procedure 2-3 times a week for 4 weeks. Study assessments will be conducted at the beginning of each week during the patient's dialysis session.
  Interventions: Device: The AquaPass System

INTERVENTIONS:
Device: The AquaPass System — The system is a non-invasive, renal-independent, single-patient, multiple-use device intended for use at the hospital, outpatient clinic, or home. The system administers warm, dry air around the patient's body to create an environmental condition that activates the eccrine glands to produce sweat, in return it removes fluids from the interstitial compartment, where fluids accumulate in fluid overload.

SUMMARY:
To demonstrate safety and performance of AquaPass System for improving fluid balance in hemo-dialysis patients, by increasing fluid loss via the skin.

DETAILED DESCRIPTION:
This study requires several investigational tests, exams, and data collection procedures to be performed by the participants. These procedures are listed in abbreviated format in the Schedule of Assessments/Activities table. The final eligibility of the trial will be confirmed after a 2-hour acclimatization session. The trial-specific procedures must not be performed until the participant has signed a written informed consent form, which has been approved by the site's Institutional Review Board.

The investigator or designee, who is trained in the clinical investigation plan, will explain the nature and scope of the trial to the participant. They will also discuss the potential risks and benefits of participation and answer any questions the participant may have. If the participant agrees to participate, they must sign the informed consent form. The investigator/designee must also sign the form before the participant can be enrolled in the trial. Any additional persons required by the site's Institutional Review Board to sign the informed consent form must also comply.

Each participant's study duration will be approximately 8 weeks. The study duration will be identical for all participants, as follows:

Screening Period: This period will last up to 7 days, during which time the participant's eligibility for the trial will be determined.

Observation Period: This period will last 3 weeks, during which the participant will come to the medical study center for weekly assessments.

Procedure Period: This period will last 4 weeks, during which time the participant will undergo 2-3 procedures with the AquaPass device each week. These procedures will be in addition to their regular hemodialysis treatment. The participant will undergo 2 procedures during the weekend, and each procedure will last 3-8 hours.

Follow-Up: This period will last 7(±1) days from the last procedure. During this period, the participant's health status will be monitored.

In summary, the study requires participants to undergo several investigational tests, exams, and data collection procedures. The study duration for each participant will be approximately 8 weeks, during which time they will undergo a screening period, observation period, procedure period, and follow-up period. All participants must provide written informed consent before any trial-specific procedures can be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Undergoing regular hemodialysis for ≥3 months
3. Subject is capable of meeting study requirements including follow-up visit
4. Subject completed 2-hour acclimatization session

Exclusion Criteria:

1. Subject is enrolled to another clinical investigation that might interfere with this study
2. Subject does not have any known skin problems (open or uncovered wounds, ulcers)
3. Subject is pregnant or planning to become pregnant within the study period, or lactating mothers
4. Scheduled living donor renal transplant during study participation
5. Has resting pre-dialysis systolic blood pressure <100mmHg
6. Limb/s amputation
7. Hyperkalemia > 6meq/d"l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Differences in weight gain over the long interdialytic period | Up to 50 days
  weight at the end of the last Hemodialysis session before AquaPass therapy subtracted from the weight in the morning of the first Hemodialysis session of the week after AquaPass therapy.
Device related Adverse Events | Up to 60 Days
  Safety evaluation of device-related adverse effects

SECONDARY OUTCOMES:
Changes in NT-proBNP | Up to 50 days
  Changes in biomarkers of congestion
Changes in Blood Urea Nitrogen | Up to 50 days
  Changes in Blood Urea Nitrogen levels
Effect on Quality of Life | up to 50 days
  change in the quality of life measured by the Kansas City Cardiomyopathy Questionnaire. In this questionnaire the minimum score is '0' and the maximum is '100', and higher scores represent a better outcome for the patient.
Affect on Ultrafiltration Rates after the long inter dialytic gap | up to 28 days
  Evaluation of the changes in ultrafiltration rates between the control phase and the Aquapass phase in the first dialysis session after the long interdialytic period

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Armaly, MD, Principal Investigator — CEO
Locations (1):
- Nazareth Hospital EMMS, Nazareth, Al Wadi Al Jawani 1611, Israel

IPD SHARING:
Plan to Share IPD: No